CLINICAL TRIAL: NCT05899400
Title: A Study to Validate and Improve an Automated Image Analysis Algorithm to Detect Tuberculosis in Sputum Smear Slides
Status: Completed | Type: Observational
Sponsor: Diascopic, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: Diascopic; 1R43EB028736-01 (NIH)
Record Dates: First submitted 2023-05-31; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Mycobacterium Sputum Slides
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: 400 Male and Female Ugandan Africans
  Interventions: Diagnostic Test: Diascopic iON Image Analysis System

INTERVENTIONS:
Diagnostic Test: Diascopic iON Image Analysis System — A scanning digital optical train that images sputum slides for automated analysis by a tuberculosis detecting algorithm

SUMMARY:
A Study to Validate and Improve an Automated Image Analysis Algorithm to Detect Tuberculosis in Sputum Smear Slides

ELIGIBILITY:
Inclusion Criteria:

* Samples sourced from Makerere University's Joint Clinical Research Clinic (JCRC) and Laboratory

Exclusion Criteria:

* No samples from outside Makerere's Domain

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 400 Male and Female Ugandan Africans
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Determined sensitivity and specificity of the iON device by comparing MTB slide results to their associated bacterial culture results from the same specimen(s). | Study completed over the grant period 2019 - 2022
  Sensitivity, specificity, and average analysis time were determined. An image database of >40,000 images was also created for internal use.

CONTACTS AND LOCATIONS:
Overall Officials: Moses Joloba, MD, PhD, Study Director — Makerere University
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No